CLINICAL TRIAL: NCT05900271
Title: Higher, Faster, Better: Is an Accelerated Intermittent Theta Burst Stimulation Protocol Compared to Standard 10 Hz Repetitive Transcranial Magnetic Stimulation, More (Cost-) Effective in Patients With Treatment-resistant Depression?
Brief Title: Dutch-Depression Outcome Trial Comparing 5 Day Multi Daily Neuronavigated Theta Burst Sessions With 6 Weeks rTMS
Acronym: DDOTT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Radboud University Medical Center (Other); Maastricht University Medical Center (Other); Maastricht University (Other); Trimbos (Unknown); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Donders Centre for Neuroscience (Other)
Responsible Party: Principal Investigator, Annemiek Dols, MD, PhD, psychiatrist and researcher, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10390012110079
Record Dates: First submitted 2023-05-10; First posted 2023-06-12 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Treatment Resistant Depression
Keywords: TMS; treatment resistant depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Intervention Model Description: multicentre, two-phase, randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: Those carrying out clinical assessments will be blinded. However, participants and those who will be administering the rTMS or SNT treatment will not be blinded. Participants and research staff will be requested not to reveal information about treatment allocation to the raters.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intermittent theta burst transcranial magnetic stimulation (iTBS) (Experimental): 5-day multi daily neuronavigated intermittent theta burst sessions (developed by Stanford University) and coined, SNT, i.e., Stanford NeuromdulaTion protocol
  Interventions: Device: iTBS
- 10 Hz repetitive-transcranial-magnetic-stimulation (rTMS) (Active Comparator): 6-weeks standard 10 Hz rTMS
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — 10 Hz repetitive-transcranial-magnetic-stimulation
  Arms: 10 Hz repetitive-transcranial-magnetic-stimulation (rTMS)
Device: iTBS — neuronavigated intermittent theta burst transcranial-magnetic-stimulation
  Arms: intermittent theta burst transcranial magnetic stimulation (iTBS)

SUMMARY:
INTRODUCTION Recent findings from three small studies (total n=59) suggest that three changes in repetitive Transcranial Magnetic Stimulation (rTMS) protocols, called the Stanford Neuromodulation Therapy (SNT) protocol, contribute to extreme high overall remission of 79% in patients with treatment resistant depression (TRD), whereas remission using a standard 10 Hz rTMS protocol is 25%. The improvement using the SNT protocol is achieved by combining 1) accelerated treatment with multiple sessions per day, 2) applying a higher overall pulse dose of stimulation, using intermittent Theta Burst Stimulation (iTBS), and 3) precise targeting of the region in the left dorsolateral prefrontal cortex (DLPFC), using functional MRI guided neuronavigation.

OBJECTIVE To determine if the SNT protocol is more (cost-) effective compared to standard 10 Hz rTMS in patients with TRD, even though the number of pulses given in both protocols is equal, i.e., 90,000.

STUDY DESIGN Multicenter randomized controlled trial comparing SNT with standard 10Hz rTMS with a follow-up of 25 weeks.

STUDY POPULATION 108 Patients with TRD (no response to 2 or more evidence-based treatments).

INTERVENTION 50 sessions using the SNT protocol in 5 days. The region of the left DLPFC most anticorrelated with the subgenual anterior cingulate cortex in each participant will be targeted based on subject-specific functional resting state MRI.

COMPARISON 30 standard daily 10 Hz rTMS sessions in six weeks, targeting the left DLPFC based on standard measurement procedures of the skull.

OUTCOME MEASURES

* Remission, based on the Hamilton depression rating scale
* Cost effectiveness, based on healthcare resource use
* Quality of life and positive mental health
* Tolerability and safety
* Relapse
* Description of opportunities and difficulties with regard to implementation

SAMPLE SIZE The investigators will enrol 108 patients (α=0.05, power is 0.80) including adjustment for attrition.

COST EFFECTIVENESS ANALYSIS SNT is faster and possibly more effective than 10Hz rTMS leading to a total cost reduction of 22 million each year considering less expensive healthcare, reduced illness duration and absence from work.

TIME SCHEDULE Within 36 months, the investigators will recruit and treat 108 patients with TRD: each center will recruit 9 patients per year. After the last follow-up assessments, the investigators will finalise the study within 12 months and report the results.

DETAILED DESCRIPTION:
Rationale: Novel therapies are crucial for patients with unipolar depression since more than 33% of these patients are medication-resistant. As a consequence, there is a high burden of illness for patients with depression, leading to increased suicide rates, inability to maintain proper work and/or social role functions, and reduced quality of life. A promising novel treatment strategy is an intensive five-day course of intermittent Theta Burst Stimulation (iTBS), a form of transcranial magnetic stimulation (rTMS), which could lead to exceptionally high remission rates (79%) in patients with treatment resistant depression. However, it remains unclear whether this novel treatment strategy is more effective in depressed patients when compared to standard 10Hz rTMS (remission 30%).

Hypothesis: 5-day multi daily neuronavigated iTBS sessions (developed by Stanford University and coined, SNT, i.e., Stanford NeuromdulaTion protocol) are more (cost-) effective than standard 10 Hz rTMS in patients with treatment resistant depression.

Objective: To determine remission of depression and cost effectiveness using the SNT protocol, in patients with treatment resistant depression who did not respond to two or more evidence-based treatments.

Study design: This study comprises a multicentre, two-phase, randomized clinical trial. Phase 1 comprises a randomized controlled trial. In Phase 1, participants will be assigned to one of the two active treatment conditions, and will receive either treatment using the SNT protocol (5 days of 10 sessions/day, resulting in 50 sessions in total 90000 pulses) or standard 10 Hz left sided rTMS, provided once daily during 6 weeks (30 sessions in total, 90000 pulses). Phase 2 comprises three follow-up measurements, one at 5 weeks, one at 10 weeks and one at 25 weeks after the last treatment with SNT or 10 Hz standard rTMS. Finally, participants who were allocated to standard 10 Hz rTMS will be offered SNT after the end of the study (e.g., 25 weeks after the last rTMS session). Patients allocated to SNT can obtain 10 Hz standard rTMS after SNT has been completed.

Study population: Adult patients with unipolar depression who did not respond to two or more evidence-based treatments for depression, in the current depressive episode, aged 18 years and over.

Sample size: Sample size calculations based on differences in remission suggest that a well-powered trial should consist of 108 patients (for a 2-sided test at alpha=0.05 and with power=0.80).

Intervention: 50 sessions using the SNT protocol in 5 days. The subregion of the left DLPFC most anticorrelated with the subgenual anterior cingulate cortex (sgACC) in each participant will be targeted based on patient-specific functional resting state magnetic resonance imaging .

Comparison: 30 standard daily 10 Hz rTMS sessions in six weeks, targeting the left DLPFC based on standard scalp-based measurement procedures.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Sufficient level of spoken and written Dutch;
* Ability to freely provide written informed consent;
* Current DSM-5 diagnosis of a depressive episode, ascertained by the Mini International Neuropsychiatry Interview (MINI-S).
* A Hamilton depression rating score (HDRS) of >16 points: this score will be obtained from the SIGH-ADS, a depression rating scale able to determine the HDRS score and a score for atypical depression.
* have a treatment resistant depression, defined according to the criteria of Conway, that is, lack of remission for eight consecutive weeks after two different evidence-based treatments anti-depressant medication has to be adequately dosed(7,24).
* Stable anti-depressant medication 6 weeks prior to study. Benzodiazepines may be used up to a dosage equivalent of 3.0 mg lorazepam, and can be lowered over time during the study based on clinical judgement.

Exclusion Criteria:

* - Bipolar disorder.
* Current psychotic disorder¸ including psychotic depression, assessed by treating psychiatrist.
* Suspected dementia, assessed with a dementia screening tool, i.e., the Montreal Cognitive Assessment (MOCA)(25), with a score of less than 20 points, or a clinical suspicion of dementia, or neuroimaging indication for neurodegeneration with a Fazekas > 1 and MTA >1. These cut-offs ensure exclusion of patients with (preclinical) dementia.
* Active suicidal thoughts and intent to act on it, assessed at the baseline interview and before the start of the trial. This assessment is based on the Columbia suicide severity rating scale, i.e., question 5 is answered positive "Have you started to work out or worked out the details of how to kill yourself? Do you intend to carry out this plan?" (26).
* Metallic devices implanted above the neck, assessed at the baseline interview.
* Patients diagnosed with epilepsy, by a neurologist, assessed at the baseline interview.
* Substance abuse 4 weeks prior to the study, including high dosage of benzodiazepine, a dosage equivalent higher than 3.0 mg lorazepam, assessed at the baseline interview.
* Inability to understand or comply with study requirements as judged by the investigators, assessed at the baseline interview.
* Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Remission | After 1 week.
  Clinical outcome is remission, which is defined as a score of 7 or lower on the clinician-rated HDRS-17 (17-itemHamilton Depression Rating Scale, scores 0-52 with higher score indicating worse outcome) measured one week after the last treatment session.

SECONDARY OUTCOMES:
Health-related quality of life | After 1-, 5-, 10- and 25-weeks.
  Health-related quality of life determined with the EQ 5D-5L (EuroQol 5 Dimension 5 Level, scores 5-25, with higher scores indicating worse outcome).
Self-rated depressive symptoms | After 1-, 5-, 10- and 25-weeks.
  Percentual reduction of depressive symptoms as measured with self-rated HDRS-6 (self-rated 6-item Hamilton Depression Rating Scale, scores 0-18 with higher score indicating worse outcome).
Relapse | After1-, 5-, 10- and 25-weeks.
  Relapse, at 5-, 10- and 25-weeks post-treatment. Relapse is defined as a HDRS-17 (17-item Hamilton Depression Rating Scale, scores 0-52 with higher score indicating worse outcome) total score of 15 or higher for 2 consecutive assessments separated by 5 to 15 days or hospitalization for depression
Side-effects | After 1- and 6- weeks.
  Establish tolerability of the treatment and side effects, of SNT and rTMS.
Remission | 5-, 10- and 25-weeks after the last treatment session.
  Clinical outcome is remission, which is defined as a score of 7 or lower on the clinician-rated HDRS-17 (17-item Hamilton Depression Rating Scale, scores 0-52 with higher score indicating worse outcome) measured directly after the last treatment session.

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - Radboud UMC, Nijmegen, GL
  - GGZinGeest, Amsterdam, North Holland
  - Amsterdam UMC location AMC, Amsterdam-Zuidoost, North Holland
  - Maastricht UMC, Maastricht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dols A, Biemans T, Coomans C, van Eijndhoven P, Dalhuisen I, van der Werf YD, Vriend C, Gomes ESA, Sack AT, Schuhmann T, Chaudhry M, Arns M, Walters BH, Wijnen B, Zalesky A, Cash R, Blumberger DM, Scheepstra KW, Hoogendoorn AW, van den Heuvel OA, van Exel E; D-DOTT Consortium. Comparison of 5-Day Multidaily Neuronavigated Theta-Burst Sessions With 6-Week Standard Repetitive Transcranial Magnetic Stimulation (the Dutch Depression Outcome Trial): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Aug 21;14:e70121. doi: 10.2196/70121. PMID 40840870